CLINICAL TRIAL: NCT07219563
Title: Open-label, 4-Part Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of Alnuctamab (BMS-986349/CC-93269) in Participants With Moderate to Severe Refractory Systemic Lupus Erythematosus
Brief Title: Alnuctamab for Refractory SLE (LATTE Study)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Chrisanna Dobrowolski, Senior Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-01686
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Refractory, Systemic Lupus Erythematosus (SLE); Severe Refractory Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with Lupus (Experimental): This study drug will be done by sentinel dosing (study drug given to a small number of participants to watch closely) before all the participants receive the study drug.
  Interventions: Drug: Alnuctamab

INTERVENTIONS:
Drug: Alnuctamab — The study drug will be given as an injection under the skin. For the first 9 days after the CC-93269 injection, subjects will be staying in the hospital. The goal of this study is to determine the optimal dose of CC-93269 to be safely administered to participants.
  Other Names: EM901

SUMMARY:
This study will assess the safety and preliminary efficacy of the bi-specific TCE, alnuctamab (known as BMS-986349, CC-93269, EM901), targeting BCMA in patients with moderate to severe SLE, refractory to standard-of-care treatments.

DETAILED DESCRIPTION:
The purpose of this research study is for researchers to learn if the investigational therapy called alnuctamab (known as BMS-986349, CC-93269, EM901) is safe and effective to treat refractory Systemic Lupus Erythematosus (SLE). CC-93269 is investigational, which means its safety and effectiveness have not been established and it is not approved by the U.S. Food and Drug Administration (FDA) for SLE. This will be the first study testing CC-93269 in SLE. Alnuctumab is a type of treatment known as a T cell engager. It is a special protein engineered in the laboratory, which is able to attach to T cells, a type of white blood cell that can kill other cells in the body. T cells normally protect the body from infections, for example by destroying the cells where the virus hides. In this case, alnuctumab will redirect T cells to a new target, called the plasma B cell. This is a type of white blood cell that plays an important role in activating the autoimmune response in patients with lupus. By linking T cells to the autoimmune plasma B cells, alnuctumab will allow the removal of these pathogenic cells. The goal is to evaluate whether this will be sufficient and safe to treat lupus.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 18-60 years.
* Documented diagnosis of SLE fulfilling 2019 ACR/EULAR criteria.
* Historical documentation of ANA (1:80 or greater) autoantibody on immunofluorescence as well as presence of at least 1 additional autoantibody of the type: anti-dsDNA, anti-histone, anti-chromatin, anti-Smith, anti-RNP, anti-Ro/SSA, anti-La/SSB, anti-cardiolipin (IgG), or anti-beta2-glycoprotein1 (IgG).
* History of SLE that is refractory to corticosteroids and at least 2 immunosuppressive therapies with different mechanisms of action (methotrexate, thiopurines, mycophenolate mofetil, calcineurin inhibitors, biologic agents, cyclophosphamide), including at least one biologic therapy (e.g. anti-CD20 therapy, anifrolumab, belimumab) or cyclophosphamide. Of note, hydroxychloroquine is not considered an immunosuppressive therapy, and methotrexate/azathioprine counts as a single drug class).
* Total SLEDAI-2K >6 with clinical SLEDAI-2K >4, or >1 BILAG A organ domain score, or >2 BILAG B, but without active central nervous system (CNS) disease within the past year; a maximum of two participants with only arthritis and/or rash can be included if truly disabling

Key Exclusion Criteria:

* Autoimmune disease other than SLE, except associated Sjogren's Disease if not primary contributor to symptoms; coexistent fibromyalgia will be allowed if not primary contributor to symptoms.
* TTP-like SLE; catastrophic APS; LN WHO class V as primary qualifying criterion (unless overlap with Class III or IV), rapidly progressive LN, or eGFR <40 mL/min; active CNS pathology attributable to neuropsychiatric SLE.
* Active or suspected infection, including HIV.
* O2 sat <92% on room air; ANC <1500u/L, Hgb <8g/dL, Plt <75,000/uL; ALT or AST > 2X ULN (unless attributed to active myositis), Total Bilirubin >1.5 X ULN (unless Gilbert's Disease), total B cell count <12/microliter, hypogammaglobinemia <500mg/dL.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of treatment emergent AEs | 9 days
  Type, frequency, and severity of treatment emergent AEs, SAEs, DLTs, and AEs of special interest (e.g., CRS, ICANS)

SECONDARY OUTCOMES:
Maximum concentration of Alnuctamab | 0-29 days
  The maximum concentration of Alnuctamab (Cmax) following multiple subcutaneous (SC) administrations in participants with moderate to severe SLE refractory to standard therapy
Change in SLE Responder Index (SRI) rate | Baseline, Week 24 and Week 52
  SLE Responder Index (SRI) rate at Week 24, Week 52 compared to baseline
  SRI is defined as the proportion of participants achieving ≥4 point reduction in SLEDAI-2K [Systemic Lupus Erythematosus Disease Activity Index], with no new A organ domain score, ≤ 1 new BILAG [British Isles Lupus Assessment Group] B score, and no worsening of the Physician Global Assessment (PGA) score
  SLEDAI-2K: Total score ranges from 0-105 with higher score indicating greater disease activity BILAG: B Score implies need for a modest dose of steroids. PGA: Score range from -3 (poorer health outcome) to 3 (better health outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Chrisanna Dobrowolski, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai School
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. For individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link tbd).